CLINICAL TRIAL: NCT00703820
Title: AML08: A Phase II Randomized Trial of Clofarabine Plus Cytarabine Versus Conventional Induction Therapy And A Phase II Study Of Natural Killer Cell Transplantation In Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Clofarabine Plus Cytarabine Versus Conventional Induction Therapy And A Study Of NK Cell Transplantation In Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML08; R01CA138744 (NIH); R01CA115422 (NIH); R01CA132946 (NIH); NCI-2011-03659 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Etoposide; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ADE (Active Comparator): Cytarabine + Daunorubicin + Etoposide
  NK cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Etoposide; Device: CliniMACS
- Clo/AraC (Active Comparator): Clofarabine + Cytarabine
  NK cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Cytarabine; Drug: Clofarabine; Device: CliniMACS

INTERVENTIONS:
Drug: Cytarabine — See Detailed Description
  Other Names: Ara-C; Cytosar-U®
Drug: Daunorubicin — See Detailed Description
  Other Names: Daunomycin; Cerubidine®
  Arms: ADE
Drug: Etoposide — See Detailed Description
  Other Names: VP-16; Vepesid®
  Arms: ADE
Drug: Clofarabine — See Detailed Description
  Other Names: Clolar^TM; Clofarex
  Arms: Clo/AraC
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System

SUMMARY:
The purpose of this study is to assess the feasibility and efficacy of a novel form of therapy-haploidentical NK cell transplantation-in patients with standard-risk AML. In addition, we will investigate the efficacy of clofarabine + cytarabine (Clo/AraC) in newly diagnosed patients with AML and attempt to optimize outcome through the use of MRD-adapted therapy and further improvements in supportive care.

DETAILED DESCRIPTION:
The overall objective of this protocol is to improve the cure rate of acute myeloid leukemia (AML).

We will compare the immunologic complete response rate after one course of therapy in patients who receive cytarabine + daunorubicin + etoposide (ADE) with that in patients who receive clofarabine + cytarabine (Clo/AraC)

Secondary objectives include

* To estimate the event-free survival (EFS) of standard risk (SR) patients who receive chemotherapy alone and the EFS of SR patients who receive chemotherapy followed by natural killer (NK) cell transplantation.

Exploratory Objectives:

* To genotype natural killer (NK) cell receptors and measure their expressions at diagnosis and after induction therapy, and to explore the associations of these features with treatment outcome
* To assess the prognostic value of levels of minimal residual disease in peripheral blood at day 8 of induction I
* To validate new markers and methods for minimal residual disease (MRD) detection
* To identify new prognostic factors by applying new technologies to study patient material
* To identify pharmacogenetic, pharmacokinetic and pharmacodynamic predictors for treatment-related outcomes in the context of the systemic therapy used in the protocol
* To describe the impact of antibiotic and antifungal prophylaxis on invasive bacterial and fungal infections, febrile neutropenia, hospitalization, and antibiotic resistance.
* To determine the performance characteristics of broad-range, molecular diagnostic methods for detection of bacterial, fungal, and viral agents, in comparison to methods currently in routine clinical use

Treatment will be based on cytogenetic and molecular characteristics, morphology, and response to therapy as assessed by flow cytometry. Risk groups are defined below. The general treatment plan will consist of chemotherapy for LR patients, chemotherapy ± NK cell therapy for SR patients, and chemotherapy + stem cell transplant (SCT) for HR patients. HR patients who do not have a suitable stem cell donor or who decline SCT will be eligible for NK cell therapy.

Low-risk (LR) criteria (not eligible for SCT or NK cell therapy)

* Core binding factor (CBF) leukemia [t(8;21)/AML1-ETO or inv(16)/t(16;16)/CBF-MYH11,] and MRD < 0.1% at day 22,regardless of other genetic features.
* Patients with CBF leukemia who have MRD ≥ to 0.1% at day 22 or who have increasing levels of fusion transcript will be considered SR and thus eligible for NK cell therapy.

Standard-risk (SR) criteria (eligible for NK cell therapy)

* Absence of low-risk or high-risk features.
* CBF leukemia with MRD ≥ 0.1% at day 22 or increasing levels of fusion transcript
* FLT3-ITD and MRD < 0.1% at day 22

High-risk (HR) criteria (candidates for SCT; eligible for NK cell therapy)

Presence of one of the following features:

* t(6;9), t(8;16), t(16;21), -7, -5, or 5q-
* FAB M0 or M6
* FAB M7 without t(1;22)
* Treatment-related (secondary) AML
* RAEB-2 or AML arising from prior MDS
* FLT3-ITD and MRD ≥ 0.1% at day 22
* All other patients with poor response to therapy (must have one of the following features) MRD ≥ to 5% at day 22 MRD ≥ to 0.1% after Induction II

Induction therapy (2 courses)

All patients will receive two courses of induction therapy that will include one course of either high dose cytarabine, daunorubicin, and etoposide (HD-ADE) or one course of clofarabine and cytarabine (Clo/AraC), followed by one course of low dose cytarabine, daunorubicin, and etoposide (LD-ADE). Patients will be randomly assigned to receive one of the following induction regimens.

Induction I: HD-ADE

Cytarabine: 3 g/m2 IV over 3 hours q12 hours x 6 doses (days 1, 3, 5) Daunorubicin: 50 mg/m2 (1.67 mg/kg for patients less than 10 kg) IV over 6 hours on days 2, 4, 6 (3 doses) Etoposide: 100 mg/m2 IV over 4 hours on days 2-6 (5 doses)

Induction I: Clo/AraC

Clofarabine: 52 mg/m2 IV over 2 hours on days 1-5 (5 doses) Cytarabine: 1 gram/m2 IV over 2 hours on days 1-5 (5 doses; each dose to start 4 hours after the start of clofarabine)

Induction II: LD-ADE

Cytarabine: 100 mg/m2 IV over 30 minutes q12 hours on days 1-8 (16 doses), Daunorubicin: 50 mg/m2 (1.67 mg/kg for patients less than 10 kg) IV over 6 hours on days 2, 4, 6 (3 doses) Etoposide: 100 mg/m2 IV over 4 hours on days 1-5 (5 doses)

Induction II for patients with FLT3-ITD: LD-ADE + Sorafenib

Patients with FLT3-ITD will take Sorafenib, 400 mg/m2 per day, orally in two divided doses (200 mg/m2/dose BID) starting one day after the completion of Induction II and continuing for 21 days Patients with FLT3-ITD who do not experience toxicity related to Sorafenib will also receive a 21-day course of Sorafenib after subsequent courses of chemotherapy.

Induction II for other HR patients: LD-ADE + vorinostat

[NOTE: Collaborating institutions may elect to opt out of treatment with vorinostat. If a site opts out, then all applicable patients at that site will receive standard induction therapy with LD-ADE (without vorinostat).]

Patients with M7 AML without t(1;22) and other HR patients without FLT3-ITD will be treated with a combination of vorinostat and LD-ADE. Vorinostat will be given orally for 3 days (Days -2, -1, 0) prior to the initiation of Induction II chemotherapy.

Special subgroup HR patients with MRD < 0.1% may proceed directly to SCT after Induction I if a suitable donor is available and the transplant can be performed without delay.

Consolidation I:

Mitoxantrone: 12 mg/m2 (0.4 mg/kg for patients less than 10 kg) IV over 1 hour on days 3-5 (3 doses) Cytarabine: 1 g/m2 IV over 2 hours every 12 hours on days 1-4 (8 doses)

Consolidation II:

Cytarabine 3 g/m2 IV over 3 hours every 12 hours on days 1, 2, 8, 9 (8 doses). Erwinia Asparaginase 25,000 Units/m2 (833 Units/kg for infants < 1 month of age, or for infants < 3 months of age who were born significantly prematurely defined as < 36 weeks gestation) IM or IV over 1 hour, 3 hours after the 4th and 8th doses of cytarabine.

NK cell therapy Standard risk patients who have a KIR-mismatched family member who is greater than 18 years old will undergo NK cell transplantation. In addition, HR patients who do not have a suitable stem cell donor or who decline SCT will be eligible for NK cell therapy if they have a KIR-mismatched family member.

Treatment schema Day -7: Cyclophosphamide 60 mg/kg IV over 1 hour. Mesna 15 mg/kg/dose IV Days -6 through -2: Fludarabine 25 mg/m2/day IV over 30 minutes (5 doses) Days -1, +1, +3, +5, +7, +9: IL-2 1 million units/m2 given subcutaneously Day -1: Donor pheresis Day 0: NK cell infusion

No steroids, including the use of hydrocortisone as pre-medication, may be given to patients during the 3 days prior to the NK cell infusion or during the first 7 days after the infusion.

CNS therapy

Triple intrathecal therapy with methotrexate, hydrocortisone, and cytarabine (MHA) will be used for all CNS therapy at the doses:

< 1 year methotrexate 6 mg, hydrocortisone 12 mg, cytarabine 18 mg, 1-2 years methotrexate 8 mg, hydrocortisone 16 mg, cytarabine 24 mg, 2-3 years methotrexate 10 mg, hydrocortisone 20 mg, cytarabine 30 mg, > 3 years methotrexate 12 mg, hydrocortisone 24 mg, cytarabine 36 mg

Leucovorin rescue (5 mg/m2 per dose; 5 mg maximum per dose) will be given orally or intravenously at 24 and 30 hours after each IT MHA treatment.

Patients with no evidence of CNS disease \[(i.e., no leukemic blast cells on cerebrospinal fluid (CSF) cytospin] will receive 4 total doses of intrathecal therapy, given at approximately one month intervals or at the beginning of each of the first 4 courses of chemotherapy.IT therapy will not be given before NK cell therapy.

Patients with overt CNS leukemia (less than or equal to 5 leukocytes per l of CSF and the presence of leukemic blast cells on CSF cytospin) will receive weekly intrathecal therapy until the CSF is free of blast cells (minimum number of doses, 4). These patients will then receive 4 additional doses of intrathecal therapy (minimum total number of doses, 8) at approximately 1-month intervals (generally given with each subsequent course of chemotherapy).IT therapy will not be given before NK cell therapy.

Patients with < 5 leukocytes per mul of CSF and the presence of leukemic blast cells on CSF cytospin (CNS2)will receive weekly intrathecal therapy until the CSF is free of blast cells. These patients will then receive 4 additional doses of intrathecal therapy at approximately 1-month intervals (generally given with each subsequent course of chemotherapy).IT therapy will not be given before NK cell therapy.

Patients who are unable to undergo lumbar puncture and receive intrathecal therapy prior to starting induction I should be treated as CNS2 unless they have overt CNS leukemia (CNS3).

ELIGIBILITY:
Inclusion Criteria:

* Age less than or equal to 21 years at time of study entry.
* No prior therapy for this malignancy except for one dose of intrathecal therapy and the use of hydroxyurea or low-dose cytarabine (100-200 mg/m2 per day for one week or less ) for hyperleukocytosis.
* Written informed consent according to institutional guidelines
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female participants must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Down syndrome
* Acute Promyelocytic Leukemia (APL)
* Juvenile Myelomonocytic Leukemia (JMML)
* Fanconi anemia (FA)
* Kostmann syndrome
* Shwachman syndrome
* Other bone marrow failure syndromes
* Use of concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of IT therapy, hydroxyurea, or low-dose cytarabine as stated above. The patient must have recovered from all acute toxicities from any previous therapy.
* Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 324 (Actual)
Dates: Start 2008-08-04 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rubnitz, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (7):
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute and Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook's Children's Medical Center, Fort Worth, Texas
- National University Health System, Singapore, Singapore

REFERENCES:
- [Derived] Rubnitz JE, Lacayo NJ, Inaba H, Heym K, Ribeiro RC, Taub J, McNeer J, Degar B, Schiff D, Yeoh AE, Coustan-Smith E, Wang L, Triplett B, Raimondi SC, Klco J, Choi J, Pounds S, Pui CH. Clofarabine Can Replace Anthracyclines and Etoposide in Remission Induction Therapy for Childhood Acute Myeloid Leukemia: The AML08 Multicenter, Randomized Phase III Trial. J Clin Oncol. 2019 Aug 10;37(23):2072-2081. doi: 10.1200/JCO.19.00327. Epub 2019 Jun 27. PMID 31246522
- [Derived] Nguyen R, Wu H, Pounds S, Inaba H, Ribeiro RC, Cullins D, Rooney B, Bell T, Lacayo NJ, Heym K, Degar B, Schiff D, Janssen WE, Triplett B, Pui CH, Leung W, Rubnitz JE. A phase II clinical trial of adoptive transfer of haploidentical natural killer cells for consolidation therapy of pediatric acute myeloid leukemia. J Immunother Cancer. 2019 Mar 20;7(1):81. doi: 10.1186/s40425-019-0564-6. PMID 30894213
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 324 participants enrolled between August 2008 and March 2017.
Pre-assignment Details: Prior to starting the study, 62 participants were excluded for the following reasons: 29 participants were donors, 8 were determined to be ineligible (wrong diagnosis), 2 were MPAL (mixed AML) patients, and 23 were not randomized.
Groups:
- Cytarabine+Daunorubicin+Etoposide: Participants receive Cytarabine + Daunorubicin + Etoposide as their first course of chemotherapy. Subsequent therapy is risk-adapted.
- Clofarabine+Cytarabine: Participants receive Clofarabine + Cytarabine as their first course of chemotherapy. Subsequent therapy is risk-adapted.
Period: Overall Study
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine
Started | 133 | 129
Completed ("For purposes of this report, a living subject *completes* the study three years after completion of therapy and the study is considered *complete* when all participants have died, been taken off study, or completed the study.") | 98 | 95
Not Completed | 35 | 34
Not completed — Adverse Event | 12 | 17
Not completed — Death | 5 | 0
Not completed — Lack of Efficacy | 11 | 11
Not completed — Received non-protocol therapy | 1 | 0
Not completed — Physician Decision | 4 | 5
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cytarabine+Daunorubicin+Etoposide: Participants receive Cytarabine + Daunorubicin + Etoposide as a first course followed by risk-adapted therapy.
- Clofarabine+Cytarabine: Participants receive Clofarabine + Cytarabine as a first course followed by risk-adapted therapy.
- Total: Total of all reporting groups
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine | Total
Number analyzed (Participants) | 133 | 129 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.57 (6.00) | 9.05 (6.40) | 9.31 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 119
  Male | 73 | 70 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 17 | 45
  Not Hispanic or Latino | 99 | 110 | 209
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 12 | 18
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 20 | 21 | 41
  White | 100 | 81 | 181
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Day 22 Minimal Residual Disease (MRD) Measured by Flow Cytometry
Description: MRD-negative is defined as <0.1% blasts with leukemia-associated phenotype detected by flow cytometry. MRD-positive is defined as >=0.1% blasts with leukemia-associated phenotype detected by flow cytometry.
Time Frame: Day 22 MRD measurement after one course of therapy
Population: Of 262 randomized patients, 242 patients were included in day 22 MRD analysis. 20 patients were excluded due to: 16 were not evaluable by flow cytometry, 2 died prior to completing the first course of therapy, 2 were off therapy for unacceptable toxicity prior to completion of one course.
Measure: Count of Participants; unit: Participants
Groups:
- Cytarabine+Daunorubicin+Etoposide: Patients received Cytarabine + Daunorubicin + Etoposide as their first course of chemotherapy. Subsequent therapy is risk-adapted.
- Clofarabine+Cytarabine: Patients received Clofarabine + Cytarabine as their first course of chemotherapy. Subsequent therapy is risk-adapted.
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine
Number analyzed (Participants) | 121 | 121
Participants
  MRD Positive | 42 | 57
  MRD Negative | 79 | 64
Statistical Analysis 1: Comparison: Cytarabine+Daunorubicin+Etoposide vs Clofarabine+Cytarabine; The study was designed to test the null hypothesis that Cytarabine+Daunorubicin+Etoposide and Clofarabine+Cytarabine result in the same proportion of patients with positive MRD after 22 days. Power calculations indicate that enrollment of a total of 240 MRD-evaluable patients in a 5-stage Haybittle-Peto group sequential design gives 80% power at the 5% level to detect an odds ratio of 2.5. The design was developed using East statistical software; Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.0429 so that the overall level of the study is maintained at 0.05 across the 4 interim analyses and the final analysis; The p-value was computed using an exact, risk-group stratified, two-sided test; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.03 to 3.41] — The odds ratio is defined as the ratio of the odds that a Clofarabine+Cytarabine patient is MRD positive to the odds that a Cytarabine+Daunorubicin+Etoposide patient is MRD positive

2. Secondary Outcome: Event-free Survival of Standard Risk Patients Who Receive Chemotherapy Alone.
Description: Kaplan-Meier estimate of the probability of being alive and free of relapse or second malignancy three years after protocol enrollment
Time Frame: 3 years after completion of therapy
Population: Randomized standard risk patients who received chemotherapy only
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Clofarabine+Cytarabine: Patients received Clofarabine + Cytarabine as their first course of chemotherapy. Subsequent therapy is risk- adapted.
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine
Number analyzed (Participants) | 51 | 41
Percentage of participants | 55.6 [43.3 to 71.4] | 54.3 [40.6 to 72.5]

3. Secondary Outcome: Event-free Survival of Standard Risk Patients Who Receive Chemotherapy Followed by Natural Killer Cell Transplantation.
Description: as for outcome 2
Time Frame: 3 years after completion of therapy
Population: Randomized patients who received NK cell therapy after chemotherapy
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine
Number analyzed (Participants) | 9 | 9
Percentage of participants | 55.6 [31.0 to 99.7] | 77.8 [54.9 to 100.0]

ADVERSE EVENTS:
Time Frame: Participants were monitored from the start of therapy through 30 days after this protocol's treatment plan was completed. Participants who received NK cell infusions were followed until any identified toxicities resolved to less than grade 2. Donors were followed for adverse events from the day of apheresis through seven days following apheresis.
Groups:
- Cytarabine+Daunorubicin+Etoposide: Participants received Cytarabine + Daunorubicin + Etoposide as their first course of chemotherapy. Subsequent therapy is risk-adapted.
- Clofarabine+Cytarabine: Participants received Clofarabine + Cytarabine as their first course of chemotherapy. Subsequent therapy is risk-adapted.
- Stem Cell Donors: This group enrolled in the study to provide donor cells to participants. Donors did not receive therapy.
Arm/Group | Cytarabine+Daunorubicin+Etoposide | Clofarabine+Cytarabine | Stem Cell Donors
All-Cause Mortality (participants affected / at risk) | 43/133 | 32/129 | 0/29
Serious Adverse Events (participants affected / at risk) | 127/133 | 122/129 | 0/29
Other Adverse Events (participants affected / at risk) | 9/133 | 9/129 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytarabine+Daunorubicin+Etoposide (N=133) | Clofarabine+Cytarabine (N=129) | Stem Cell Donors (N=29)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 33 (47) | 48 (62) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 45 (78) | 48 (90) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 20 (26) | 27 (35) | 0 (0)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 4 (5) | 4 (4) | 0 (0)
Allbumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7 (10) | 4 (6) | 0 (0)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 7 (7) | 11 (15) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 16 (19) | 14 (15) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 (8) | 8 (10) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 16 (20) | 14 (16) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 11 (12) | 13 (18) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Potassium, serum-ghigh (hyperkalemia) (Metabolism and nutrition disorders) | 2 (3) | 5 (9) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 17 (22) | 10 (14) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 7 (7) | 7 (7) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fibrinogen (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (11) | 15 (19) | 0 (0)
Pain, throat/pharynx/larynx (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Mucositis/stomatitis (clinical exam), oral cavity (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 14 (17) | 0 (0)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 6 (6) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 16 (18) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 5 (5) | 0 (0)
Hemorrhage, GI, Oral cavity (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
Pain, Abdomen NOS (Gastrointestinal disorders) | 4 (6) | 5 (6) | 0 (0)
Pain, Anus (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstruction, GI, Sotmach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage, GI, Lower GI NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Pain, rectum (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Perforation, GI, appendix (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pain, oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, abdomen NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pain, stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam), small bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucotitis/stomatitis (functional/symptomatic), esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, lip (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0)
Pain, head/headache (Nervous system disorders) | 4 (4) | 3 (5) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy: cranial, CN VI lateral deviation of eye (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
CNS necrosis/cystic progression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurology - other (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy: cranial, CN IX Motor-pharynx; sensory-ear, pharynx, tongue (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Infection (documented clinically or microbiologically documented, ANC<1.0x10e9/L, fever>38.5C),blood (Infections and infestations) | 20 (23) | 21 (24) | 0 (0)
Infection (documented clinically or microbioogically) with Grade 3 or 4 neutrophils (ANC<1.0x10e9/L) (Infections and infestations) | 71 (103) | 77 (115) | 0 (0)
Infection - other (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 7 (7) | 15 (16) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 21 (25) | 18 (18) | 0 (0)
Infection with unknown ANC, blood (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Infection with unknown ANC, lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC, urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC, catheter-related (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection with unknown ANC, lip/perioral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 11 (13) | 8 (8) | 0 (0)
Allergy/immunology - other (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction to Asparaginase (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (fever of unknown origin: not clinically or microbiologically documented) (Blood and lymphatic system disorders) | 90 (189) | 95 (194) | 0 (0) — ANC <1.0x10e9/L, fever >=38.5C
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular/visual - other (Eye disorders) | 0 (0) | 0 (0) | 0 (0)
Ocular surface disease (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic disc edema (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Death not associated with CTCAE term, multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Constitutional symptoms - other (General disorders) | 1 (2) | 2 (3) | 0 (0)
Weight loss (General disorders) | 3 (4) | 3 (5) | 0 (0)
Injection site reaction/extravasation changes (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain - other (General disorders) | 1 (2) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0x10e9/L) (General disorders) | 10 (10) | 6 (6) | 0 (0)
Edema: head and neck (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death not associated with CTCAE term, sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 19 (20) | 0 (0)
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Hemorrhage, pulmonary/upper respiratory, nose (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory, bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Valvular heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrhythmia - other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
Cardiac general - other (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 3 (4) | 2 (2) | 0 (0)
Supraventricular and nodal arrhythmia, sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Right ventricular dysfunction (cor pulmonale) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia, sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain, skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/bleeding - other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (12) | 5 (5) | 0 (0)
Hypotension (Vascular disorders) | 8 (9) | 9 (9) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Hematoma (Vascular disorders) | 3 (4) | 0 (0) | 0 (0)
Pain, back (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain, extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Pain, buttock (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain, joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Growth and development - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, chest wall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy), extremity-upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Investigations) | 2 (2) | 4 (4) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1 (1) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (4) | 3 (3) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/genitourinary - other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
Incontinence, urinary (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Mood alteration, anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood alteration, depression (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Personality/behavioral (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood alteration, agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood alteration, euphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Intra-operative injury - other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatobiliary/pancreas - other (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pain, vagina (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GU, iuterus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytarabine+Daunorubicin+Etoposide (N=133) | Clofarabine+Cytarabine (N=129) | Stem Cell Donors (N=29)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 9 (11) | 9 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT00703820/Prot_SAP_001.pdf